CLINICAL TRIAL: NCT00325689
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, 16 Week Study of Aripiprazole Used as Dual Therapy in the Treatment of Patients With Chronic Stable Schizophrenia or Schizoaffective Disorder Demonstrating an Inadequate Response to Quetiapine or Risperidone Monotherapy.
Brief Title: Aripiprazole Used as Dual Therapy in the Treatement of Patients With Chronic Stable Schizophrenia or Schizoaffective Disorder.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-397 ST
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2011-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Quetiapine Fumarate; Risperidone; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Quetiapine or Risperidone + Aripiprazole (Active Comparator)
  Interventions: Drug: Quetiapine or Risperidone + Aripiprazole
- Quetiapine or Risperidone + placebo (Placebo Comparator)
  Interventions: Drug: Quetiapine or Risperidone + placebo

INTERVENTIONS:
Drug: Quetiapine or Risperidone + Aripiprazole — Tablets, Oral, Quetiapine 400-800 mg/day or Risperidone (4-8 mg/day) + Aripiprazole 2-15 mg/day, Flexible, 16 weeks.
  Other Names: Abilify
  Arms: Quetiapine or Risperidone + Aripiprazole
Drug: Quetiapine or Risperidone + placebo — Tablets, Oral, Quetiapine 400-800 mg/day or Risperidone (4-8 mg/day) + Placebo, Flexible, 16 weeks.
  Arms: Quetiapine or Risperidone + placebo

SUMMARY:
A Multicenter, Double-blind 16 Week Study on the augmentation of atypical antipsychotic with Aripiprazole in patients with Schizophrenia with inadequate response to antipsychotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of chronic Schizophrenia or Schizoaffective disorder
* Stable symptoms and dose of Quetiapine or Risperidone

Exclusion Criteria:

* First diagnosis in the past year
* Significant risk of suicide or meet DSM-IV-TR criteria for substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of adding Aripiprazole to atypical antipsychotic treatment via Positive and Negative Symptoms Scale (PANSS) score at endpoint | (Week 16) or at time of discontinuation

SECONDARY OUTCOMES:
Assess efficacy according to changes in the severity of illness symptoms as measured by the Clinical Global Impressions-Severity (CGI-S) | at endpoint (Week 16)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (48):
- United States (48):
  - K & S Professional Research Services, Llc, Little Rock, Arkansas
  - Comprehensive Neuroscience, Inc., Cerritos, California
  - Atp Clinical Research, Inc., Costa Mesa, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - San Fernando Mental Health Center, Granada Hills, California
  - Uci Medical Center, Orange, California
  - California Clinical Trials Medical Group, Paramount, California
  - California Clinical Trials, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - California Neuropsychopharmacology Clinical Research Inst., San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Department Of Psychiatry And Behavioral Sciences, Stanford, California
  - Pacific Clinical Research Medical Group, Upland, California
  - University Of Colorado At Denver And Health Sciences Center, Denver, Colorado
  - Institute Of Living, Hartford, Connecticut
  - Behavioral Clinical Research, Inc, North Miami, Florida
  - Uptown Research Institute, Llc, Chicago, Illinois
  - Alexian Center For Psychiatric Research, Hoffman Estates, Illinois
  - Indiana University School Of Medicine, Indianapolis, Indiana
  - Lsu Health Sciences Center, Shreveport, Louisiana
  - J. Gary Booker, Md, Shreveport, Louisiana
  - Sheppard Pratt Health System, Baltimore, Maryland
  - North Suffolk Mental Health Association, Boston, Massachusetts
  - Community Counseling Of Bristol County, Inc. (Ccbc), Taunton, Massachusetts
  - University Of Minnesota, Minneapolis, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - Cri Worldwide, Llc, Clementon, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Advanced Bio-Behavioral Sciences, Elmsford, New York
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - New York State Psychiatric Institute, New York, New York
  - Manhattan Psychiatric Center, New York, New York
  - Strong Ties Community Support Program, Rochester, New York
  - Behavioral Medical Research Of Staten Island, Staten Island, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Duke University Health System, Durham, North Carolina
  - Saroj B. Brar, M.D., Inc., Cleveland, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Department Of Veterans Affairs Medical Center, Coatesville, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Va Medical Center (116a), Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Belmont Center For Comprehensive Treatment, Philadelphia, Pennsylvania
  - Cri Worldwide, Llc, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Medlabs Research Of Houston, Inc., Houston, Texas
  - University Of Texas Health Science Center At San Antonio, San Antonio, Texas
  - Va Puget Sound Health Care System, Tacoma, Washington

REFERENCES:
- [Background] Kane JM, Correll CU, Goff DC, Kirkpatrick B, Marder SR, Vester-Blokland E, Sun W, Carson WH, Pikalov A, Assuncao-Talbott S. A multicenter, randomized, double-blind, placebo-controlled, 16-week study of adjunctive aripiprazole for schizophrenia or schizoaffective disorder inadequately treated with quetiapine or risperidone monotherapy. J Clin Psychiatry. 2009 Oct;70(10):1348-57. doi: 10.4088/JCP.09m05154yel. PMID 19906340